CLINICAL TRIAL: NCT04783194
Title: Dexamethasone Plus Bupivacaine Versus Bupivacaine in Bilateral Trans-incisional Paravertebral Block in Lumbar Spine Surgeries, a Randomized Clinical Trial.
Brief Title: Dexamethasone Plus Bupivacaine Versus Bupivacaine in Bilateral Trans-incisional Paravertebral Block in Lumbar Spine Surgeries .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 47/2020/2021
Record Dates: First submitted 2021-02-28; First posted 2021-03-05 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone + bupivacaine in bilateral TiPVB in lumbar spine surgery (Active Comparator): Dexamethasone plus bupivacaine in bilateral trans-incisional paravertebral block in lumbar spine surgery for postoperative analgesia
  Interventions: Drug: Dexamethasone+ Bupivacaine
- Bupivacaine in bilateral TiPVB in lumbar spine surgery (Active Comparator): Bupivacaine in bilateral trans-incisional paravertebral block in lumbar spine surgery for postoperative analgesia
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone+ Bupivacaine — Dexamethasone plus bupivacaine in bilateral trans-incisional paravertebral block in lumbar spine surgery.
  Arms: Dexamethasone + bupivacaine in bilateral TiPVB in lumbar spine surgery
Drug: Bupivacaine — Bupivacaine in bilateral trans-incisional paravertebral block in lumbar spine surgery.
  Arms: Bupivacaine in bilateral TiPVB in lumbar spine surgery

SUMMARY:
The purpose of this study is to compare addition of dexamethasone to bupivacaine versus bupivacaine alone for trans-incisional bilateral paravertebral block for postoperative analgesia in elective lumbar spine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* physical status American Society of Anesthesiologists (ASA) I or II.

Exclusion Criteria:

* refuse to participate have a body mass index (BMI) >30 kg/m2 ASA physical status >II have major illnesses (e.g., cardiac, respiratory, renal, hepatic or neurological) coagulation abnormalities infection at the injection site tumor in the paravertebral space sepsis Severe chest deformity or scoliosis, due to the possibility of injection into the meninges an allergy or contraindications to the drugs used in the study uncontrolled diabetes patients with active gastric ulceration a history of drug addiction or alcohol abuse a psychiatric illness mental retardation interfering with the evaluation of pain scores.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | 1st 24 hour
  After extubation, an IV PCA system will be connected to the patient (Accufuser Plus® 100 mL: Woo Young Medical Co, Korea). PCA will be prepared with 60 mL of normal saline containing 60 mg of morphine, and the system will be programmed to give a 0.5 mL bolus dose with a lockout interval of 8 min. basal rate will not be present. PCA will be discontinued at 24 h after surgery, and at that time, oral analgesics begin.

SECONDARY OUTCOMES:
Total opioid consumption . | 1st 24 hour
  Total opioid consumption in the first 24 h postoperatively .
Visual analogue scale (VAS) | 1st 24 hours postoperatively
  Pain scores will be evaluated by a blinded observer anesthesiologist at the time of arrival in the PACU and 10, 20, and 30 min and 1, 2, 4, 6, 12, and 24 h thereafter using a visual analog scale (VAS) (ranging from0-10 cm: where 0 = no pain, 10 = worst pain). The patients Will be instructed about the usage of the PCA system and the VAS preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt